CLINICAL TRIAL: NCT01936792
Title: Pathology in the Brain After mTBI - A Multimodal MRI Study
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Hammel Neurocenter (Other)
Responsible Party: Principal Investigator, Erhard Trillingsgaard Næss-Schmidt, Pathology in the brain after mTBI - A multimodal MRI study, University of Aarhus
Other Study IDs: 1-10-72-135-13
Record Dates: First submitted 2013-08-21; First posted 2013-09-06 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-03

CONDITIONS: Concussion
Keywords: Concussion; Mild Traumatic Brain Injury; Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- mild traumatic brain injury: Subjects with mild traumatic brain injury
- Controls: Controls with no premorbid health conditions

SUMMARY:
The purpose is to use Diffusion Kurtosis Imaging (DKI), Diffusion Tensor Imaging (DTI) and resting state functional MRI to examine tissue damage in the brains of people who have had a concussion, both acute and 3 months after the accident. A secondary purpose is to examine whether the results of the scans are associated with physical, cognitive and emotional problems after concussion.

It is hypothesized that there will be a change in the diffusion signal measured with DKI in the thalamus (THA) and with DTI in the corpus callosum (CC), in the acute stage and at follow-up of the mTBI subjects compared with the healthy controls. Secondary it is expected that there will be changes in the diffusion signal measured with DKI and DTI in other WM and GM area in both the acute stage and at follow up with mTBI subjects compared with healthy controls. Also rs-fMRI markers are secondary expected to differ in the two groups. Moreover secondarily the MRI markers are tested for correlation with the severity of PCS acutely and at follow up after mTBI.

DETAILED DESCRIPTION:
More than 25,000 people in Denmark, are each year diagnosed with commotio cerebri as a result of head trauma (National Patient Registry, 1996), and foreign studies report that up to 5 to 15% of these have symptoms that persist beyond 3 months (5). Post commotio symptoms (PCS) are typically divided into physical, cognitive and emotional symptoms and include headache, fatigue, memory loss, stress, etc.. It is known from previous studies of traumatic brain injuries that the cost of the disabling process and the failure to intervene in the long term are very costly (11). In Denmark there are to date no systematic or consistent treatment for people with persistent symptoms 3 months after commotio cerebri, and a lack of general knowledge about the pathology and standardization with regard to diagnosis and prognosis are also missing.

Commotio cerebri, also known as mild traumatic brain injury (mTBI) is often defined as an exogenous traumatic stimulus that causes a physiological disruption of brain function (American Congress of Rehabilitation Medicine). This includes a biochemical cascade, edema, micro-haemorrhages, diffuse axonal injury (DAI) and changes in activity between internal networks in the brain (12, 13).

In severe trauma, conventional scanning methods such as Computer Tomography (CT) and Magnetic Resonance Imaging (MRI) can detect bone rupture, edema and micro-haemorrhages, but in mTBI, it is often difficult to detect edema or micro-hemorrhages, and the conventional methods is often not sensitive enough to show pathology especially beyond the acute period, although patients continue to have physical symptoms as well as cognitive and emotional problems (6, 12).

More MRI techniques, which are not routinely used in the clinic, has verified both DAI and changes in cortical network as compared to healthy controls (12). One of these is the method Diffusional tensor imaging (DTI) which can be used to detect the DAI in white matter (WM). DTI studies confirm DAI in several WM areas after mTBI (12). Other studies have shown that DAI detected by DTI in several places of WM correlates with cognitive problems after mTBI (1,2,6,13).

A more recent and less studied MRI method is Diffusional Kurtosis Imaging (DKI) which can display DAI in WM and prove to be more sensitive than the DTI for the detection of damage in gray matter (GM) (3, 4). A study in humans showed significant differences between individuals with mTBI and healthy controls, in the thalamus and several WM areas (3). This study also showed a correlation between DKI markers in the thalamus and the capsula interna with cognitive problems in multiple domains after mTBI. DKI is therefore suggested to be used in addition to DTI in relation to detect tissue damage in both WM and GM.

Another MRI method that has shown promising results in relation to mTBI is resting state functional MRI (fMRI-rs). Rs-fMRI has shown differences between brain network connectivity in mTBI patients compared to healthy controls (9). A study based on the theory Default Mode Network (DMN) has also shown a high degree of sensitivity and specificity in a patient classification in the subacute phase (8).

Generally more longitudinal studies, larger publications with more participants and consensus on which areas that are associated with MRI verified pathology are still missing. Also the correlations between MRI markers with the physical, cognitive and emotional problems are still to be solved.

It is the purpose to use three research based scan methods to detect tissue damage in the brains of persons after concussion, both acute and 3 months after the accident. Moreover the correlation between MRI makers and the registered physical, cognitive and emotional symptoms after concussion are to be examined.

It is hypothesized that there will be a change in Mean Kurtosis in the thalamus, corpus callosum and hippo campus from baseline to follow-up. Secondary we examine change in Mean Diffusivity and Fractional Anisotropy in the thalamus, corpus callosum and hippo campus from baseline to follow-up and for both DKI and DTI we examine the difference between the mTBI subjects and healthy controls in the acute stage and at follow-up. Moreover we examine correlation of MRI markers the severity of PCS acutely and at follow up. Finally rs-fMRI and default mode network is expected to differ between the two groups

Materials and methods

The study design is a controlled observational trial with follow up. 35 individuals with mTBI and 35 matched healthy controls (age and sex) are examined. Persons with mTBI are scanned within the first 14 days after mTBI and at follow-up 3 months after. Controls are scanned only once.

The MRI scans will be performed on CE-approved MRI scanners at Aarhus University Hospital, Noerrebrogade 44, 8000 Aarhus C, Denmark. A standard protocol for MRI will be used containing a structural T1, a susceptibility weighted image (SWI) and T2 FLAIR sequence with the purpose to visualize anatomy, micro hemorrhages and edema. It is expected that the findings from the standard protocol will be present in the acute stage but only for some at follow-up.

The novelty of the current study is the use of a optimized and newly developed faster DKI scan sequence, which makes it possible to use DKI in a clinical setup. In addition, to date there has not been provided a follow-up at 3 months after mTBI with DKI (9 months Grossman study).

Symptom Questionnaires:

Both at baseline and at 3 months follow-up three questionnaires are to be filled out "The Rivermead postconcussion symptom questionnaire", " The Symptom Checklist" (SCL-8AD) and The Brief Illness Perception questionnaire" (BIPQ). Control Persons will also fill out these questionnaires.

Statistical considerations:

Power calculations of the upcoming study is based upon a previous studies by Grossman et. al.(3) MK in THA at Baseline: 35 mTBI subjects (mean 0.74, sd 0.08), 35 healthy controls (mean 0.89, sd 0.04), power = 100% MK in THA at Follow up: 25 mTBI (mean 0.78, sd 0.06), 25 healthy controls (mean 0.89, sd 0.12) power = 96% An ANOVA will be used to test the difference in signal to the two times (<14 days and 3 months after mTBI).

Additionally, there will be made paired comparison between mTBI individuals. Both primary and secondary outcomes will showed in uncorrected and Bonferroni corrected.

Regions and parameters which show significant differences, will be compared with symptom scores using Spearman rank correlation, controlled for age and sex.

Risks, side effects and disadvantages:

MRI:

All project participants will review a checklist compared with contraindications for. There is no evidence of harmful effects of MRI, if these precautions are followed. Additionally subjects are provided with earplugs to protect from the noise from the scanner.

The clinical scans will be seen by a neuroradiologist and if abnormality is suspected, pictures will be evaluated further. If the abnormality is real the subject will get an additional examine and appropriate guidance will be conducted by the involved neuroradiologist.

While the images from the research part is not primarily used for clinical use, there will not be made any clinical diagnostic evaluation from these brain scans and they are not necessarily evaluated by a person with clinical radiological competence.

Research Ethics statement:

The techniques used are non-invasive and does not include methods like intravascular catheters, injection of contrast agents or any medication. There is no radiation danger, and the studies are not associated with significant side effects, risks or disadvantages for the participants.

The project involves only competent subjects participating voluntarily after adequate verbal and written information and written consent. The participation may at any time leave the study and the investigation without having to justify it. The study itself does not involve treatment and if the subject withdraws his agreement, this does not affect his right to present or future treatment

Recruitment:

People with concussions will be recruited from the Department of Radiology at Aarhus University Hospital. Controls are recruited in the recruitment system Sona Systems and by posters with contact information.

Notification to the Data Protection Agency:

The project is registered to the data inspectorate in Region Midtjylland's of "Health Scientific research in Central Denmark Region". Personal information will be kept confidential and will be destroyed after the study is completed. The project is progressing in accordance with the Act on Processing of Personal Data (http://www.datatilsynet.dk/borger/forskningsprojekter/).

Publication of results:

Publication of results from the project will be coordinated by the Project Manager in accordance with the guidelines specified in the "Guidelines for Good Scientific Practice" (Committee on Scientific Dishonesty, 1998).

Positive as well as negative, and results that can not be concluded on, will be published in international scientific journals.

Financial support:

The project is initiated by the Hospital of Hammel Neuro Center. There is no sponsorship or secondary economic interests involved in the project.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-40 years
* negative CT scan
* A Glasgow Coma Scale (GCS) score that is higher than 13 after 30 minutes
* one or more of the following characteristics:
* A period of loss of consciousness for up to 30 minutes
* A period of amnesia of events immediately before or after the accident within 24 hours before / after the episode
* Any change in mental state at the time of the accident (eg, dazed, disoriented or confused)
* Focal neurological deficit, which may or may not be transient

Exclusion Criteria:

* Psychiatric or neurological diagnosis already
* The use of drugs, smoking or alcohol eight hours before MRI
* Alcohol or drug abuse
* Former mTBI with unconsciousness within the last 2 years
* Significant other trauma, as the primary symptom
* MRI contraindications

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 35 individuals with mTBI and 35 matched healthy controls (age and sex) are examined.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in Mean Kurtosis (MK) in mTBI subjects | from baseline within 14 days and to follow up 3 month after mTBI
  MRI measurement unit

SECONDARY OUTCOMES:
Difference in MK between mTBI and control subjects | within 14 days and 3 month after mTBI
  MRI measurement unit
Difference in Fractional Anisotropy (FA) between mTBI and control subjects | within 14 days and 3 month after mTBI
  MRI measurement unit
Difference in Mean Diffusivity (MD) between mTBI and control subjects | within 14 days and 3 month after mTBI
  MRI measurement unit
Change of FA in mTBI subjects | from baseline within 14 days and to follow up 3 month after mTBI
  MRI measurement unit
Change of MD in mTBI subjects | from baseline within 14 days and to follow up 3 month after mTBI
  MRI measurement unit
Correlation of clinical symptoms and MRI measurements | within 14 days and 3 month after mTBI
  questionnaire and MRI measurement units
Default mode network | within 14 days and 3 month after mTBI
  measuring the default mode network with resting state -fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen F Nielsen, Professor, Study Chair — Region Hospital, Hammel Neurocenter, University Clinic, Voldbyvej 15, 8450 Hammel
Locations (1):
- Region Hospital Hammel Neurocenter, Hammel, Denmark

REFERENCES:
- [Background] Aoki Y, Inokuchi R, Gunshin M, Yahagi N, Suwa H. Diffusion tensor imaging studies of mild traumatic brain injury: a meta-analysis. J Neurol Neurosurg Psychiatry. 2012 Sep;83(9):870-6. doi: 10.1136/jnnp-2012-302742. Epub 2012 Jul 14. PMID 22797288
- [Background] Beauchamp MH, Ditchfield M, Babl FE, Kean M, Catroppa C, Yeates KO, Anderson V. Detecting traumatic brain lesions in children: CT versus MRI versus susceptibility weighted imaging (SWI). J Neurotrauma. 2011 Jun;28(6):915-27. doi: 10.1089/neu.2010.1712. Epub 2011 Jun 9. PMID 21501069
- [Background] Grossman EJ, Ge Y, Jensen JH, Babb JS, Miles L, Reaume J, Silver JM, Grossman RI, Inglese M. Thalamus and cognitive impairment in mild traumatic brain injury: a diffusional kurtosis imaging study. J Neurotrauma. 2012 Sep;29(13):2318-27. doi: 10.1089/neu.2011.1763. Epub 2011 Sep 15. PMID 21639753
- [Background] Grossman EJ, Jensen JH, Babb JS, Chen Q, Tabesh A, Fieremans E, Xia D, Inglese M, Grossman RI. Cognitive impairment in mild traumatic brain injury: a longitudinal diffusional kurtosis and perfusion imaging study. AJNR Am J Neuroradiol. 2013 May;34(5):951-7, S1-3. doi: 10.3174/ajnr.A3358. Epub 2012 Nov 22. PMID 23179649
- [Background] Iverson GL. Outcome from mild traumatic brain injury. Curr Opin Psychiatry. 2005 May;18(3):301-17. doi: 10.1097/01.yco.0000165601.29047.ae. PMID 16639155
- [Background] Jeter CB, Hergenroeder GW, Hylin MJ, Redell JB, Moore AN, Dash PK. Biomarkers for the diagnosis and prognosis of mild traumatic brain injury/concussion. J Neurotrauma. 2013 Apr 15;30(8):657-70. doi: 10.1089/neu.2012.2439. PMID 23062081
- [Background] Lovden M, Bodammer NC, Kuhn S, Kaufmann J, Schutze H, Tempelmann C, Heinze HJ, Duzel E, Schmiedek F, Lindenberger U. Experience-dependent plasticity of white-matter microstructure extends into old age. Neuropsychologia. 2010 Nov;48(13):3878-83. doi: 10.1016/j.neuropsychologia.2010.08.026. Epub 2010 Sep 15. PMID 20816877
- [Background] Mayer AR, Mannell MV, Ling J, Gasparovic C, Yeo RA. Functional connectivity in mild traumatic brain injury. Hum Brain Mapp. 2011 Nov;32(11):1825-35. doi: 10.1002/hbm.21151. Epub 2011 Jan 21. PMID 21259381
- [Background] McDonald BC, Saykin AJ, McAllister TW. Functional MRI of mild traumatic brain injury (mTBI): progress and perspectives from the first decade of studies. Brain Imaging Behav. 2012 Jun;6(2):193-207. doi: 10.1007/s11682-012-9173-4. PMID 22618832
- [Background] Messe A, Caplain S, Paradot G, Garrigue D, Mineo JF, Soto Ares G, Ducreux D, Vignaud F, Rozec G, Desal H, Pelegrini-Issac M, Montreuil M, Benali H, Lehericy S. Diffusion tensor imaging and white matter lesions at the subacute stage in mild traumatic brain injury with persistent neurobehavioral impairment. Hum Brain Mapp. 2011 Jun;32(6):999-1011. doi: 10.1002/hbm.21092. Epub 2010 Jul 28. PMID 20669166
- [Background] PALLESEN, H. and TRIER, M., eds, 2006. Inde i varmen eller ude på et sidespor. En redegørrelse om unge med erhvervet hjerneskade og deres særlige problemstillinger. First edn. Denmark: Videnscenter for Hjerneskade.
- [Background] Toledo E, Lebel A, Becerra L, Minster A, Linnman C, Maleki N, Dodick DW, Borsook D. The young brain and concussion: imaging as a biomarker for diagnosis and prognosis. Neurosci Biobehav Rev. 2012 Jul;36(6):1510-31. doi: 10.1016/j.neubiorev.2012.03.007. Epub 2012 Mar 28. PMID 22476089
- [Background] Vagnozzi R, Signoretti S, Cristofori L, Alessandrini F, Floris R, Isgro E, Ria A, Marziali S, Zoccatelli G, Tavazzi B, Del Bolgia F, Sorge R, Broglio SP, McIntosh TK, Lazzarino G. Assessment of metabolic brain damage and recovery following mild traumatic brain injury: a multicentre, proton magnetic resonance spectroscopic study in concussed patients. Brain. 2010 Nov;133(11):3232-42. doi: 10.1093/brain/awq200. Epub 2010 Aug 23. PMID 20736189
- [Background] Voelbel GT, Genova HM, Chiaravalotti ND, Hoptman MJ. Diffusion tensor imaging of traumatic brain injury review: implications for neurorehabilitation. NeuroRehabilitation. 2012;31(3):281-93. doi: 10.3233/NRE-2012-0796. PMID 23093455